CLINICAL TRIAL: NCT00841568
Title: A Long-term Administration Study of OPC-41061 in Patients With Autosomal Dominant Polycystic Kidney Disease (ADPKD) [Extension of Study 156-04-001]
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Kyoji Imaoka, Operating Officer, Director, Department of Clinical Research and Development, Otsuka Pharmaceutical Co., Ltd.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 156-05-002; JapicCTI-090690
Record Dates: First submitted 2009-02-09; First posted 2009-02-11 (Estimated); Results first posted 2018-07-27 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: ADPKD; Tolvaptan
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: OPC-41061

INTERVENTIONS:
Drug: OPC-41061 — orally administered at 15 mg twice daily (morning and evening) for a maximum of 3 years.

SUMMARY:
Investigation into the long-term safety and efficacy of OPC-41061 in repeated oral administrations at doses of 15 mg twice daily in patients with ADPKD who completed the preceding dose-finding study (156-04-001).

DETAILED DESCRIPTION:
Investigation into the long-term safety and efficacy of OPC-41061 in repeated oral administrations at doses of 15 mg twice daily in patients with ADPKD who completed the preceding dose-finding study (156-04-001).

ELIGIBILITY:
Inclusion Criteria:

* Patients who completed 5-day repeated administrations and the follow-up observation in the preceding study (156-04-001)
* Patients in whom the safety of repeated administration was confirmed based on the investigator's reports from the preceding study (156-04-001)

Exclusion Criteria:

* Patients with serum creatinine concentration of 2.5 mg/dL or higher at the screening examination
* Patients with any of the following complications

  * Uncontrolled hypertension
  * Serious cardiovascular disease (eg. heart failure) or hepatic disease (eg. cirrhosis)"
* Patients with any of the following complications or history thereof

  * Clinically significant drug allergies (anaphylaxis) or hypersensitivity (especially, hypersensitivity to benzazepine derivatives or suspected hypersensitivity thereto)
  * Inability to personally give consent due to a mental disease "
* Patients with SBP (in sitting position) <90 mm Hg (at screening examination)
* Patients with history of massive bleeding or bleeding tendency
* Patients with a history of drug or alcohol abuse within 6 months prior to the screening examination
* Pregnant women, lactating women, or women who may become or plan to become pregnant
* Patients who received any investigational drug other than OPC-41061 within 30 days prior to commencement of administration of OPC-41061
* Any patient who, in the opinion of the principle investigator or attending investigators, should not participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-04; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kanto Region, Japan

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039
- [Derived] Higashihara E, Torres VE, Chapman AB, Grantham JJ, Bae K, Watnick TJ, Horie S, Nutahara K, Ouyang J, Krasa HB, Czerwiec FS; TEMPOFormula and 156-05-002 Study Investigators. Tolvaptan in autosomal dominant polycystic kidney disease: three years' experience. Clin J Am Soc Nephrol. 2011 Oct;6(10):2499-507. doi: 10.2215/CJN.03530411. Epub 2011 Sep 8. PMID 21903984

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OPC-41061
Started | 17
Completed | 12
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2
Not completed — Creatinine over the withdrawal criteria | 1

BASELINE CHARACTERISTICS:
Arm/Group | OPC-41061
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.8 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 8
Region of Enrollment [Number; unit: participants]
  Japan | 17

OUTCOME MEASURES:

1. Primary Outcome: Total Kidney Volume
Description: Individual subject data on the volumes of the total kidney volume (sum of the volumes of the left and right kidneys) measured by magnetic resonance imaging or computed tomography during trial period.
  Number of participants analyzed at each time point represents number of participants with data at the specified time point. Patients who were withdrawn from trial or have no appropriate data (e.g., interruption of medication, protocol deviation, etc.) are excluded.
Time Frame: Baseline, week 24, 52, 104, and 156
Measure: Median (Inter-Quartile Range); unit: mL
Groups:
- Baseline; Week 24; Week 52; Week 104; Week 156: Orally administered at 15 mg twice daily (morning and evening) for a maximum of 3 years.
  Individual subject data on the volumes of the total kidney volume (sum of the volumes of the left and right kidneys) measured by magnetic resonance imaging or computed tomography during trial period.
Arm/Group | Baseline | Week 24 | Week 52 | Week 104 | Week 156
Number analyzed (Participants) | 17 | 15 | 14 | 12 | 9
mL | 1500.5 [781.5 to 5060.1] | 1573.1 [770.0 to 5036.6] | 1567.9 [774.2 to 4940.3] | 1729.4 [858.4 to 4869.0] | 1647.7 [868.0 to 2563.8]

2. Primary Outcome: Renal Function Test (eGFR)
Description: Individual subject data on eGFR (estimated glomerular filtration rate calculated by Japanese eGFR equation) during trial period.
  Number of participants analyzed at each time point represents number of participants with data at the specified time point. Patients who were withdrawn from trial or have no appropriate data (e.g., interruption of medication, protocol deviation, etc.) are excluded.
Time Frame: Baseline, Week 24, 48, 104, and 156
Measure: Median (Inter-Quartile Range); unit: mL/min/1.73m2
Arm/Group | Baseline | Week 24 | Week 52 | Week 104 | Week 156
Number analyzed (Participants) | 17 | 15 | 14 | 12 | 12
mL/min/1.73m2 | 63.0 [33 to 108] | 64.0 [29 to 115] | 64.0 [35 to 122] | 58.5 [35 to 114] | 59.0 [27 to 103]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | OPC-41061
All-Cause Mortality (participants affected / at risk) | 1/17
Serious Adverse Events (participants affected / at risk) | 2/17
Other Adverse Events (participants affected / at risk) | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-41061 (N=17)
Diverticulitis (Infections and infestations) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OPC-41061 (N=17)
Anaemia (Blood and lymphatic system disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 3
Sinus bradycardia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 3
Asthenopia (Eye disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Keratitis (Eye disorders) | 2
Eye pruritus (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 2
Enterocolitis (Gastrointestinal disorders) | 1
Gastric polyps (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 3
Gastritis erosive (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Periodontal disease (Gastrointestinal disorders) | 1
Periodontitis (Gastrointestinal disorders) | 1
Gastrointestinal telangiectasia (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Fatigue (General disorders) | 1
Malaise (General disorders) | 2
Mass (General disorders) | 1
Oedema peripheral (General disorders) | 1
Thirst (General disorders) | 9
Inflammation (General disorders) | 1
Vessel puncture site haematoma (General disorders) | 1
Anaphylactic reaction (Immune system disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Acute tonsillitis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 13
Paronychia (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Tinea pedis (Infections and infestations) | 2
Tonsillitis (Infections and infestations) | 1
Urethritis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Arthropod sting (Injury, poisoning and procedural complications) | 2
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Laceration (Injury, poisoning and procedural complications) | 1
Muscle injury (Injury, poisoning and procedural complications) | 1
Tooth injury (Injury, poisoning and procedural complications) | 1
Mouth injury (Injury, poisoning and procedural complications) | 1
Muscle strain (Injury, poisoning and procedural complications) | 2
Contusion (Injury, poisoning and procedural complications) | 6
Wound (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Blood antidiuretic hormone increased (Investigations) | 5
Blood calcium increased (Investigations) | 1
Blood cholesterol increased (Investigations) | 2
Blood creatine phosphokinase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 2
Blood glucose increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 1
Blood osmolarity decreased (Investigations) | 1
Blood osmolarity increased (Investigations) | 1
Blood triglycerides increased (Investigations) | 2
Blood uric acid increased (Investigations) | 4
Gamma-glutamyltransferase increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 1
Monocyte count increased (Investigations) | 1
Neutrophil count increased (Investigations) | 1
Red blood cell count decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Blood phosphorus increased (Investigations) | 2
Blood alkaline phosphatase decreased (Investigations) | 1
Urine output increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Amnesia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Glossopharyngeal neuralgia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Hyperaesthesia (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Intracranial aneurysm (Nervous system disorders) | 2
Migraine (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Subarachnoid haemorrhage (Nervous system disorders) | 1
Arachnoid cyst (Nervous system disorders) | 1
Adjustment disorder with depressed mood (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Nocturia (Renal and urinary disorders) | 2
Pollakiuria (Renal and urinary disorders) | 2
Polyuria (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Breast cyst (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dyshidrosis (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No